CLINICAL TRIAL: NCT01260714
Title: A Phase I Study of Azacitidine Combined With Mitoxantrone and Etoposide (A-NOVE) Chemotherapy for Patients' Age ≥ 60 With Poor Prognosis Acute Myeloid Leukemia (AML)
Brief Title: Azacitidine, Mitoxantrone Hydrochloride, and Etoposide in Treating Older Patients With Poor-Prognosis Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate accrual rate
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02559; NCI-2011-02559 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000690647; PHL-074 (Other: University Health Network-Princess Margaret Hospital); 8331 (Other: CTEP); N01CM00032 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-06

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia; Adult Acute Monoblastic Leukemia; Adult Acute Monocytic Leukemia; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With Maturation; Adult Acute Myeloid Leukemia With Minimal Differentiation; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); RUNX1-RUNX1T1; Adult Acute Myeloid Leukemia With t(9;11)(p22;q23); MLLT3-MLL; Adult Acute Myeloid Leukemia Without Maturation; Adult Acute Myelomonocytic Leukemia; Adult Erythroleukemia; Adult Pure Erythroid Leukemia; Alkylating Agent-Related Acute Myeloid Leukemia; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Erythroblastic, Acute | interventions — Azacitidine; Etoposide; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (azacitidine, mitoxantrone hydrochloride, etoposide) (Experimental): Patients receive induction therapy comprising azacitidine SC QD on days 1-7, mitoxantrone hydrochloride IV over 30 minutes, and etoposide IV over 1 hour on days 4-8. Patients may receive up to 2 additional courses of the same treatment as re-induction or consolidation therapy beginning 35-60 days from the start of the previous course.
  Interventions: Drug: Azacitidine; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: Azacitidine — Given SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan

SUMMARY:
This phase I trial studies the best dose of azacitidine and to see how well it works with mitoxantrone hydrochloride and etoposide in treating older patients with acute myeloid leukemia that has a lower chance of responding to treatment or higher risk of returning (poor prognosis). Drugs used in chemotherapy, such as azacitidine, mitoxantrone hydrochloride, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the highest tolerated dose of two dosing schedules of azacitidine when combined with mitoxantrone (mitoxantrone hydrochloride) and etoposide (A-NOVE) chemotherapy in poor prognosis older patients with acute myeloid leukemia (AML).

II. To evaluate the toxicity of this regimen.

SECONDARY OBJECTIVES:

I. To determine the complete response (CR) rate and using this regimen. II. To evaluate changes in topoisomerase II activity, deoxyribonucleic acid (DNA) methylation and DNA expression arrays in leukemia cells during azacitidine treatment, and to correlate these changes with responses to A-NOVE chemotherapy.

III. To evaluate relapse-free survival (RFS) and overall survival (OS) in patients receiving post-remission consolidation with A-NOVE in patients achieving CR. (OS follow-up discontinued as of 08/07/2014)

OUTLINE: This is a dose-escalation study of azacitidine.

Patients receive induction therapy comprising azacitidine subcutaneously (SC) once daily (QD) on days 1-7, mitoxantrone hydrochloride IV over 30 minutes, and etoposide IV over 1 hour on days 4-8. Patients may receive up to 2 additional courses of the same treatment as re-induction or consolidation therapy beginning 35-60 days from the start of the previous course.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Acute myeloid leukemia (AML) as defined by World Health Organization (WHO) criteria, any subtype, de novo or secondary, except acute promyelocytic leukemia (APL)
* One of the following:

  * Previously untreated, with adverse-risk cytogenetics, including any one of the following:

    * Complete or partial deletion of chromosome 7
    * Complete or partial deletion of chromosome 5
    * At least 3 numerical or structural abnormalities, other than t(15;17), t(8;21) or inv(16) or variant
    * 11q23 abnormalities
    * Inv(3) or variant such as t(3:3)
  * Previously untreated, transformed from prior myelodysplastic syndrome (MDS) or myeloproliferative disorder (MPD) other than CML
  * Persistent leukemia following one cycle of 3+7 induction therapy (cytarabine plus either daunorubicin or idarubicin), any cytogenetic risk group
* Left ventricular ejection fraction (LVEF) > 50% based on multi gated acquisition scan (MUGA) scan or 2-dimensional (2-D) echocardiogram
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Serum bilirubin =< 1.5 x ULN
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Karnofsky >= 60%)
* Patients with high initial white blood cell (WBC) should have the WBC reduced to below 50 x 10^9/L with hydroxyurea, to minimize the risk of leukostasis related-complications; hydroxyurea is permitted up to 24 hours prior to starting azacitidine
* Men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; men should not father a child while participating in this study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy or investigational agents within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who have received prior radiation greater than 3000 cGy to marrow producing areas
* Patients may not be receiving any other investigational agents
* Patients with active central nervous system (CNS) leukemia; prior CNS leukemia is permitted provided the cerebrospinal fluid has cleared and there is no other evidence of active CNS leukemia
* Prior therapy for AML with decitabine, azacitidine, mitoxantrone, or etoposide
* Prior therapy with azacitidine or decitabine for pre-existing MDS
* History of allergic reactions attributed to decitabine, azacitidine, etoposide, mitoxantrone, or compounds of similar chemical or biologic composition
* Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients with cluster of differentiation (CD) counts less than 500/mm^3 and/or a history of HIV/acquired immune deficiency syndrome (AIDS)-related complications will be excluded from the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of azacitidine that can be safely combined with mitoxantrone hydrochloride and etoposide chemotherapy | Up to 2 courses of treatment
  The descriptions and grading scales found in the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting.

SECONDARY OUTCOMES:
Changes in DNA methylation | Baseline to day 4
  Nonquantitative comparisons will be made between responders and non-responders with respect to changes in DNA methylation.
Changes in gene expression | Baseline to day 4
  Nonquantitative comparisons will be made between responders and non-responders with respect to changes in gene expression.
Changes in topoisomerase II levels | Baseline to day 4
  These will be compared between responders (i.e. those achieving either CR or morphologic leukemia-free state [MLFS]) vs. non-responders (those not achieving CR/MLFS after 1-2 induction cycles), with 95% confidence intervals and 2-tailed t-tests of significance.
Complete response rate | Up to 4 years
Overall survival | From the start of study treatment until death from any cause or last follow up, assessed up to 4 years
Relapse-free survival | From documentation of CR or MLFS to time of disease recurrence or last follow up, assessed up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Brandwein, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario